CLINICAL TRIAL: NCT05420961
Title: A Phase 3 Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-Experienced Adults 50 Years of Age or Older
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-experienced Adults (V116-006, STRIDE-6)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V116-006; jRCT2071220025 (Registry Identifier: jRCT); 2021-006679-41 (EudraCT Number)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohorts 1 and 2: participants, investigator, sponsor Cohort 3: no blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: V116 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V116 on Day 1. Participants in this arm received PPSV23 prior to the enrollment.
  Interventions: Biological: V116
- Cohort 1: PCV15 (Active Comparator): Participants will receive a single 0.5 mL IM injection of PCV15 on Day 1. Participants in this arm received PPSV23 prior to the enrollment.
  Interventions: Biological: PCV15
- Cohort 2: V116 (Experimental): Participants will receive a single 0.5 mL IM injection of V116 on Day 1. Participants in this arm received PCV13 prior to the enrollment.
  Interventions: Biological: V116
- Cohort 2: PPSV23 (Active Comparator): Participants will receive a single 0.5 mL IM injection of PPSV23 on Day 1. Participants in this arm received PCV13 prior to the enrollment.
  Interventions: Biological: PPSV23
- Cohort 3: V116 (Experimental): Participants will receive a single 0.5 mL IM injection of V116 on Day 1. Participants in this arm received PCV15, PCV20, PCV13+PPSV23, PCV15+PPSV23, or PPSV23+PCV13 prior to the enrollment.
  Interventions: Biological: V116

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 4 μg of each of the pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: Cohort 1: V116; Cohort 2: V116; Cohort 3: V116
Biological: PCV15 — Pneumococcal 15-valent conjugate vaccine with 2 μg of each of the PnPs antigen: 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F, and 4 μg of 6B in each 0.5 mL sterile suspension
  Other Names: VAXNEUVANCE™
  Arms: Cohort 1: PCV15
Biological: PPSV23 — Pneumococcal 23-valent vaccine with 25 μg of each of the PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PNEUMOVAX™23
  Arms: Cohort 2: PPSV23

SUMMARY:
This a study of V116 in adults ≥50 years of age who previously received a pneumococcal vaccination ≥1 year before enrollment. The primary objectives of this study are to evaluate the safety, tolerability, and immunogenicity of V116.

DETAILED DESCRIPTION:
Participants will be randomized to 1 of 3 cohorts depending upon prior vaccinations. Prior vaccinations by cohort include: PPSV23 (pneumococcal vaccine, polyvalent [23-valent], PNEUMOVAX™23) for Cohort 1; PCV13 (pneumococcal 13-valent conjugate vaccine; PREVNAR 13™) for Cohort 2; PCV15 (pneumococcal 15-valent conjugate vaccine; VAXNEUVANCE™), PCV20 (pneumococcal 20-valent conjugate vaccine; PREVNAR 20™), PCV13+PPSV23, PCV15+PPSV23, or PPSV23+PCV13 for Cohort 3.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has received pneumococcal vaccine >= 1 year before enrollment (PCV13, PCV15, PCV20, PPSV23, PCV13+PPSV23, PPSV23+PCV13, or PCV15+PPSV23).

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD).
* Has a known hypersensitivity to any component of V116, PCV15, PCV20, or PPSV23, including diphtheria toxoid.
* Has a known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease.
* Has a coagulation disorder contraindicating intramuscular vaccination.
* Has a known malignancy that is progressing or has required active treatment.
* Has received PPSV23 followed by either PCV15 or PCV20.
* Received systemic corticosteroids (prednisone equivalent of ≥20 mg/day).
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease.
* Has received any non-live vaccine ≤14 days before receipt of study vaccine or is scheduled to receive any non-live vaccine ≤30 days after receipt of any study vaccine.
* Has received any live virus vaccine ≤30 days before receipt of study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of study vaccine.
* Has received a blood transfusion or blood products, including immunoglobulin ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product until the Day 30 post-vaccination blood draw is complete.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (51):
- United States (15):
  - Central Research Associates ( Site 0024), Birmingham, Alabama
  - Lenzmeier Family Medicine/CCT Research ( Site 0008), Glendale, Arizona
  - Fiel Family and Sports Medicine, PC/CCT Research ( Site 0006), Tempe, Arizona
  - Southland Clinical Research Center ( Site 0026), Fountain Valley, California
  - Diablo Clinical Research, Inc. ( Site 0019), Walnut Creek, California
  - Alliance for Multispecialty Research, LLC ( Site 0020), Coral Gables, Florida
  - Indago Research & Health Center, Inc ( Site 0005), Hialeah, Florida
  - Advanced Medical Research Institute ( Site 0018), Miami, Florida
  - Solaris Clinical Research ( Site 0025), Meridian, Idaho
  - Centennial Medical Group ( Site 0002), Elkridge, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division ( Site 0016), Troy, Michigan
  - Meridian Clinical Research, LLC ( Site 0009), Norfolk, Nebraska
  - Advanced Medical Research ( Site 0001), Maumee, Ohio
  - University of Texas Medical Branch-Sealy Institute for Vaccine Sciences Clinical Trials Program ( Si, Galveston, Texas
  - Health Research of Hampton Roads, Inc. ( Site 0003), Newport News, Virginia
- Canada (5):
  - Hamilton Medical Research Group ( Site 0114), Hamilton, Ontario
  - Milestone Research Inc. ( Site 0104), London, Ontario
  - Manna Research Mirabel ( Site 0109), Mirabel, Quebec
  - CHU de Québec-Université Laval-Équipe de recherche en vaccination ( Site 0120), Québec, Quebec
  - Diex Recherche Sherbrooke Inc. ( Site 0101), Sherbrooke, Quebec
- France (4):
  - CHU Bordeaux Haut-Leveque ( Site 0202), Pessac, Aquitaine
  - CHRU de Brest ( Site 0200), Brest, Finistere
  - centre hospitalier lyon sud ( Site 0204), Pierre-Bénite, Rhone
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0203), Paris
- Israel (7):
  - Rambam Health Care Campus ( Site 0303), Haifa
  - Maccabi Health Services - Holon ( Site 0305), Holon
  - Maccabi Healthcare Services ( Site 0306), Jerusalem
  - Hadassah Medical Center-Clinical Reaserch Unit ( Site 0300), Jerusalem
  - Meir Medical Center ( Site 0301), Kfar Saba
  - Sheba Medical Center-Early Phase Clinical Trials Unit ( Site 0304), Ramat Gan
  - Clalit Health Services - Sakhnin Community Clinic-Research Unit ( Site 0302), Sakhnin
- Italy (4):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 0400), Milan, Lombardy
  - Ospedale San Raffaele ( Site 0403), Milan, Lombardy
  - A.O.U. Policlinico Paolo Giaccone ( Site 0402), Palermo, Sicily
  - Azienda Ospedaliero Universitaria Policlinico Riuniti di Foggia ( Site 0405), Foggia
- Japan (2):
  - PS Clinic ( Site 0700), Fukuoka
  - Nishikumamoto Hospital ( Site 0701), Kumamoto
- South Korea (6):
  - Gachon University Gil Medical Center ( Site 0755), Namdong-gu, Incheon
  - Korea University Ansan Hospital ( Site 0751), Ansan-si, Kyonggi-do
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital ( Site 0752), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 0753), Seoul
  - Hallym University Kangnam Sacred Heart Hospital-Internal Medicine ( Site 0754), Seoul
  - Korea University Guro Hospital ( Site 0750), Seoul
- Spain (6):
  - HOSPITAL CLÍNIC DE BARCELONA-Medicina Preventiva i Epidemiologia ( Site 0503), Barcelona, Catalonia
  - EBA CENTELLES ( Site 0500), Centelles, Catalonia
  - Hospital Universitari de Bellvitge ( Site 0505), L'Hospitalet de Llobregat, Catalonia
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-Respiratory ( Site 0508), Pozuelo de Alarcón, Madrid
  - Hospital Internacional Xanit ( Site 0520), Benalmádena, Malaga
  - Hospital La Princesa ( Site 0515), Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital ( Site 0801), Tainan
  - National Taiwan University Hospital ( Site 0800), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Scott P, Haranaka M, Choi JH, Stacey H, Dionne M, Greenberg D, Grijalva CG, Orenstein WA, Fernsler D, Gallagher N, Zeng T, Li J, Platt HL; STRIDE-6 Study Group. A Phase 3 Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-Experienced Adults 50 Years of Age or Older (STRIDE-6). Clin Infect Dis. 2024 Dec 17;79(6):1366-1374. doi: 10.1093/cid/ciae383. PMID 39082735
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26093&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 717 adults were randomized to 1 of 3 cohorts. One participant randomized to receive PCV15 in Cohort 1 incorrectly received V116. Per protocol the participant was included in the Cohort 1 V116 group. One participant randomized to receive PCV15 in Cohort 1 incorrectly received PPSV23 (intervention for Cohort 2). Per protocol this participant was excluded from the all participants as treated population because the actual intervention received was not 1 of the 2 designated interventions in Cohort 1.
Groups:
- Cohort 1: V116: Participants received a single 0.5 mL intramuscular (IM) injection of V116 on Day 1. Participants in this arm received PPSV23 (pneumococcal vaccine, polyvalent [23-valent], PNEUMOVAX™23) prior to the enrollment.
- Cohort 1: PCV15: Participants received a single 0.5 mL IM injection of PCV15 (pneumococcal 15-valent conjugate vaccine; VAXNEUVANCE™) on Day 1. Participants in this arm received PPSV23 prior to the enrollment.
- Cohort 2: V116: Participants received a single 0.5 mL IM injection of V116 on Day 1. Participants in this arm received PCV13 (pneumococcal 13-valent conjugate vaccine; PREVNAR 13™) prior to the enrollment.
- Cohort 2: PPSV23: Participants received a single 0.5 mL IM injection of PPSV23 on Day 1. Participants in this arm received PCV13 prior to the enrollment.
- Cohort 3: V116: Participants received a single 0.5 mL IM injection of V116 on Day 1. Participants in this arm received PCV15, PCV13+PPSV23, PCV15+PPSV23, or PPSV23+PCV13 prior to the enrollment.
Period: Overall Study
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Started | 231 | 119 | 176 | 85 | 106
Day 1 - Vaccinated With V116 | 229 | 1 (This participant inadvertently received V116. Per protocol this participant was included in the Cohort 1 V116 group.) | 174 | 0 | 105
Day 1 - Vaccinated With PCV15 | 0 | 117 | 0 | 0 | 0
Day 1 - Vaccinated With PPSV23 | 0 | 1 (This participant inadvertently received PPSV23. Per protocol this participant was excluded from the all participants as treated (APaT) population because the actual intervention received was not one of the two designated interventions in Cohort 1.) | 0 | 85 | 0
Completed | 229 | 118 | 173 | 85 | 105
Not Completed | 2 | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Randomized by mistake without study treatment | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116 | Total
Number analyzed (Participants) | 231 | 119 | 176 | 85 | 106 | 717
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (7.5) | 69.0 (7.1) | 65.4 (7.8) | 65.4 (6.6) | 71.0 (7.6) | 67.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 60 | 101 | 49 | 56 | 383
  Male | 114 | 59 | 75 | 36 | 50 | 334
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 17 | 34 | 16 | 14 | 103
  Not Hispanic or Latino | 207 | 102 | 142 | 69 | 92 | 612
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 96 | 47 | 55 | 25 | 13 | 236
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 3 | 1 | 6 | 19
  White | 127 | 69 | 118 | 59 | 86 | 459
  More than one race | 2 | 0 | 0 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following any injection with either V116, PCV15, or PPSV23 the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were erythema, pain, and swelling.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 230 | 117 | 174 | 85 | 105
Percentage of Participants
  Injection site erythema | 7.4 | 7.7 | 7.5 | 9.4 | 7.6
  Injection site pain | 35.7 | 43.6 | 41.4 | 47.1 | 43.8
  Injection site swelling | 8.3 | 8.5 | 4.6 | 16.5 | 10.5

2. Primary Outcome: Percentage of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following any of the injections with either V116, PCV15, or PPSV23, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were fatigue, headache, myalgia, and pyrexia.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 230 | 117 | 174 | 85 | 105
Percentage of Participants
  Fatigue | 14.3 | 17.1 | 19.0 | 12.9 | 21.9
  Headache | 7.0 | 9.4 | 10.3 | 11.8 | 8.6
  Myalgia | 7.4 | 2.6 | 9.8 | 9.4 | 8.6
  Pyrexia | 1.7 | 2.6 | 2.9 | 1.2 | 0.0

3. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. The percentage of participants with one or more SAE that were assessed by the investigator to be at least possibly related to the study vaccination are presented.
Time Frame: Up to ~180 days
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 230 | 117 | 174 | 85 | 105
Percentage of Participants | 0.4 | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Geometric Mean Titer (GMT) of Serotype-specific Opsonophagocytic Activity (OPA)
Description: OPA for the serotypes contained in V116 were determined using a multiplex opsonophagocytic assay (MOPA). GMT is defined as geometric mean titer (1/dil). Serotype-specific OPA GMTs with 95% confidence intervals are presented.
Time Frame: 30 Days post-vaccination
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity endpoint and who had sufficient data to perform the analyses were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 215 | 115 | 166 | 78 | 99
Titers
  Serotype 3: number analyzed (Participants) | 197 | 103 | 149 | 75 | 85
  Serotype 3 | 262.1 [224.0 to 306.8] | 226.3 [182.0 to 281.4] | 391.1 [332.8 to 459.6] | 583.1 [453.5 to 749.6] | 318.3 [250.0 to 405.3]
  Serotype 6A: number analyzed (Participants) | 191 | 94 | 152 | 74 | 93
  Serotype 6A | 1653.5 [1347.2 to 2029.4] | 2076.1 [1571.4 to 2742.8] | 3624.0 [3099.2 to 4237.7] | 1812.3 [1226.6 to 2677.6] | 2097.3 [1693.4 to 2597.6]
  Serotype 7F: number analyzed (Participants) | 209 | 110 | 150 | 70 | 96
  Serotype 7F | 2184.4 [1891.4 to 2522.8] | 1750.3 [1404.7 to 2181.0] | 3129.8 [2609.9 to 3753.3] | 4057.0 [3211.2 to 5125.6] | 2051.3 [1630.2 to 2581.0]
  Serotype 19A: number analyzed (Participants) | 204 | 109 | 158 | 74 | 93
  Serotype 19A | 1513.8 [1318.4 to 1738.1] | 2022.9 [1634.1 to 2504.3] | 2528.9 [2201.7 to 2904.9] | 3241.5 [2646.0 to 3971.0] | 1533.8 [1272.4 to 1848.9]
  Serotype 22F: number analyzed (Participants) | 206 | 108 | 143 | 71 | 99
  Serotype 22F | 1983.8 [1698.3 to 2317.4] | 1595.6 [1227.1 to 2074.6] | 4389.2 [3541.1 to 5440.3] | 2524.0 [1834.5 to 3472.5] | 1913.5 [1453.5 to 2519.0]
  Serotype 33F: number analyzed (Participants) | 188 | 99 | 131 | 59 | 88
  Serotype 33F | 4311.9 [3625.1 to 5128.9] | 3397.2 [2665.3 to 4330.0] | 8162.9 [6407.2 to 10399.7] | 8761.9 [6157.4 to 12468.1] | 4654.3 [3532.1 to 6133.1]
  Serotype 8: number analyzed (Participants) | 208 | 113 | 161 | 75 | 98
  Serotype 8 | 1273.0 [1115.1 to 1453.3] | 345.8 [250.5 to 477.5] | 2320.1 [1987.3 to 2708.7] | 2723.2 [2197.4 to 3374.8] | 1486.8 [1230.5 to 1796.6]
  Serotype 9N: number analyzed (Participants) | 191 | 111 | 143 | 58 | 90
  Serotype 9N | 3805.1 [3324.0 to 4356.0] | 2176.5 [1809.6 to 2617.9] | 7214.4 [6062.9 to 8584.6] | 6482.5 [4908.9 to 8560.7] | 4054.5 [3389.4 to 4850.2]
  Serotype 10A: number analyzed (Participants) | 209 | 112 | 155 | 73 | 96
  Serotype 10A | 1986.2 [1637.7 to 2408.9] | 467.5 [337.0 to 648.5] | 3976.8 [3360.7 to 4705.8] | 1797.6 [1136.2 to 2843.9] | 2564.0 [1959.1 to 3355.6]
  Serotype 11A: number analyzed (Participants) | 197 | 100 | 142 | 71 | 87
  Serotype 11A | 1998.5 [1696.9 to 2353.8] | 335.6 [228.9 to 491.8] | 2846.6 [2411.0 to 3360.8] | 1736.6 [1367.1 to 2206.1] | 2373.0 [1905.4 to 2955.4]
  Serotype 12F: number analyzed (Participants) | 212 | 114 | 160 | 73 | 99
  Serotype 12F | 981.8 [782.4 to 1232.1] | 80.5 [54.0 to 120.1] | 2252.6 [2120.5 to 3072.9] | 1402.5 [912.2 to 2156.4] | 1235.3 [948.3 to 1609.2]
  Serotype 15A: number analyzed (Participants) | 175 | 93 | 134 | 63 | 86
  Serotype 15A | 4184.9 [3548.3 to 4935.6] | 877.2 [616.2 to 1248.7] | 6185.2 [5179.3 to 7386.6] | 1668.2 [1234.4 to 2254.5] | 4328.6 [3378.7 to 5545.7]
  Serotype 15C: number analyzed (Participants) | 206 | 110 | 152 | 72 | 89
  Serotype 15C | 2307.8 [1878.4 to 2835.4] | 539.6 [371.1 to 784.6] | 4334.4 [3563.8 to 5271.5] | 1470.4 [978.6 to 2209.3] | 2191.9 [1573.2 to 3053.9]
  Serotype 16F: number analyzed (Participants) | 187 | 107 | 146 | 74 | 89
  Serotype 16F | 3060.5 [2633.8 to 3556.3] | 392.3 [301.3 to 510.8] | 4626.5 [3861.8 to 5542.6] | 832.8 [604.3 to 1147.6] | 2477.0 [1887.2 to 3251.2]
  Serotype 17F: number analyzed (Participants) | 194 | 108 | 125 | 67 | 82
  Serotype 17F | 3599.8 [3134.5 to 4134.3] | 939.6 [693.7 to 1272.6] | 5963.8 [5036.6 to 7061.7] | 4367.3 [3372.5 to 5655.7] | 3836.7 [3063.4 to 4805.1]
  Serotype 20A: number analyzed (Participants) | 195 | 110 | 138 | 72 | 88
  Serotype 20A | 2847.4 [2433.3 to 3331.8] | 1058.9 [829.9 to 1351.1] | 6005.5 [4919.8 to 7330.8] | 3393.9 [2536.9 to 4540.5] | 2433.4 [1880.5 to 3148.9]
  Serotype 23A: number analyzed (Participants) | 202 | 91 | 156 | 60 | 86
  Serotype 23A | 2363.9 [1857.4 to 3008.5] | 310.2 [202.1 to 476.0] | 4253.4 [3417.6 to 5293.5] | 433.6 [247.5 to 759.5] | 3967.2 [2764.8 to 5692.7]
  Serotype 23B: number analyzed (Participants) | 197 | 110 | 160 | 75 | 97
  Serotype 23B | 673.2 [517.1 to 876.4] | 153.0 [98.7 to 237.1] | 1530.7 [1196.5 to 1958.3] | 203.9 [127.6 to 325.6] | 844.0 [608.2 to 1171.4]
  Serotype 24F: number analyzed (Participants) | 201 | 97 | 151 | 63 | 90
  Serotype 24F | 1822.6 [1411.6 to 2353.3] | 106.6 [69.7 to 162.9] | 2746.1 [2257.9 to 3339.9] | 48.5 [28.6 to 82.1] | 2041.5 [1500.8 to 2777.1]
  Serotype 31: number analyzed (Participants) | 194 | 108 | 146 | 68 | 90
  Serotype 31 | 3018.4 [2473.6 to 3683.3] | 113.2 [74.5 to 172.1] | 4413.5 [3530.2 to 5517.7] | 171.8 [99.9 to 295.6] | 3285.5 [2485.0 to 4343.8]
  Serotype 35B: number analyzed (Participants) | 194 | 107 | 148 | 76 | 90
  Serotype 35B | 6703.1 [5732.7 to 7837.8] | 1019.1 [739.9 to 1403.7] | 8143.5 [6761.4 to 9808.1] | 1527.7 [1169.5 to 1995.5] | 5836.8 [4693.6 to 7258.6]

5. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG)
Description: The geometric mean concentration (GMC) of serotype-specific immunoglobulin G (IgG) for the serotypes contained in V116 was determined using a pneumococcal electrochemiluminescence (PnECL) assay. Serotype-specific pneumococcal IgG GMCs with 95% confidence intervals are presented.
Time Frame: 30 Days post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 220 | 117 | 167 | 81 | 99
μg/mL
  Serotype 3 | 0.87 [0.77 to 0.99] | 0.80 [0.65 to 0.97] | 0.89 [0.77 to 1.03] | 1.58 [1.25 to 2.00] | 0.85 [0.70 to 1.03]
  Serotype 6A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 6A | 4.69 [3.72 to 5.90] | 7.69 [5.60 to 10.57] | 7.81 [6.30 to 9.68] | 5.24 [3.62 to 7.56] | 5.48 [4.27 to 7.03]
  Serotype 7F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 7F | 5.71 [4.89 to 6.68] | 6.45 [5.08 to 8.19] | 5.65 [4.75 to 6.73] | 8.34 [6.57 to 10.59] | 5.07 [4.12 to 6.23]
  Serotype 19A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 19A | 8.54 [7.33 to 9.95] | 11.97 [9.40 to 15.24] | 9.12 [7.70 to 10.81] | 12.41 [9.57 to 16.11] | 8.06 [6.50 to 9.98]
  Serotype 22F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 22F | 4.41 [3.69 to 5.28] | 4.33 [3.37 to 5.56] | 5.38 [4.34 to 6.66] | 2.87 [2.12 to 3.87] | 3.08 [2.36 to 4.01]
  Serotype 33F | 13.36 [11.22 to 15.91] | 12.72 [10.37 to 15.61] | 15.04 [12.31 to 18.37] | 13.92 [10.23 to 18.94] | 9.66 [7.53 to 12.40]
  Serotype 8 | 9.58 [8.21 to 11.17] | 3.56 [2.74 to 4.62] | 11.29 [9.28 to 13.73] | 14.47 [10.86 to 19.27] | 7.48 [5.87 to 9.53]
  Serotype 9N: number analyzed (Participants) | 217 | 117 | 167 | 81 | 99
  Serotype 9N | 7.06 [5.92 to 8.43] | 3.59 [2.83 to 4.55] | 8.48 [6.89 to 10.44] | 7.32 [5.47 to 9.78] | 4.15 [3.23 to 5.34]
  Serotype 10A | 9.86 [7.99 to 12.18] | 2.77 [2.12 to 3.63] | 18.21 [14.30 to 23.18] | 7.29 [4.94 to 10.74] | 10.03 [7.21 to 13.98]
  Serotype 11A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 11A | 7.16 [6.09 to 8.42] | 2.06 [1.65 to 2.58] | 9.13 [7.44 to 11.22] | 3.95 [2.98 to 5.23] | 4.78 [3.79 to 6.03]
  Serotype 12F | 1.46 [1.18 to 1.81] | 0.41 [0.30 to 0.55] | 1.91 [1.44 to 2.53] | 1.01 [0.65 to 1.56] | 0.96 [0.70 to 1.31]
  Serotype 15A | 16.35 [13.45 to 19.88] | 1.56 [1.19 to 2.05] | 20.24 [15.92 to 25.75] | 2.15 [1.52 to 3.03] | 11.16 [7.91 to 15.75]
  Serotype 15C: number analyzed (Participants) | 219 | 117 | 166 | 81 | 99
  Serotype 15C | 11.08 [9.01 to 13.62] | 3.25 [2.37 to 4.45] | 16.67 [12.78 to 21.76] | 4.31 [2.91 to 6.38] | 6.51 [4.72 to 8.99]
  Serotype 16F: number analyzed (Participants) | 218 | 117 | 166 | 81 | 99
  Serotype 16F | 4.69 [3.75 to 5.87] | 0.37 [0.28 to 0.48] | 4.04 [3.19 to 5.10] | 0.30 [0.22 to 0.41] | 2.46 [1.78 to 3.41]
  Serotype 17F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 17F | 13.20 [11.18 to 15.58] | 2.68 [2.08 to 3.46] | 14.96 [12.37 to 18.08] | 7.23 [5.26 to 9.92] | 9.92 [7.86 to 12.53]
  Serotype 20A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 20A | 14.83 [12.37 to 17.77] | 4.93 [3.83 to 6.36] | 22.21 [17.77 to 27.75] | 10.73 [7.48 to 15.41] | 12.16 [8.99 to 16.46]
  Serotype 23A: number analyzed (Participants) | 219 | 117 | 166 | 81 | 99
  Serotype 23A | 5.38 [4.19 to 6.90] | 0.75 [0.55 to 1.02] | 6.03 [4.55 to 7.99] | 0.62 [0.43 to 0.90] | 4.25 [2.88 to 6.26]
  Serotype 23B: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 23B | 6.66 [5.53 to 8.03] | 2.61 [1.96 to 3.48] | 6.00 [4.91 to 7.33] | 2.31 [1.75 to 3.06] | 5.05 [3.90 to 6.54]
  Serotype 24F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 24F | 10.05 [7.59 to 13.32] | 0.49 [0.39 to 0.61] | 7.48 [5.45 to 10.46] | 0.31 [0.23 to 0.42] | 6.12 [3.84 to 9.75]
  Serotype 31: number analyzed (Participants) | 217 | 117 | 167 | 81 | 99
  Serotype 31 | 4.48 [3.66 to 5.48] | 0.37 [0.30 to 0.47] | 3.58 [2.87 to 4.46] | 0.32 [0.24 to 0.44] | 3.66 [2.64 to 5.08]
  Serotype 35B: number analyzed (Participants) | 218 | 117 | 167 | 81 | 99
  Serotype 35B | 26.31 [21.60 to 32.04] | 1.45 [1.18 to 1.78] | 24.55 [20.09 to 30.01] | 1.45 [1.17 to 1.80] | 18.15 [13.61 to 24.21]

6. Secondary Outcome: Geometric Mean Fold Rise in Serotype-specific Opsonophagocytic Activity (OPA)
Description: Activity for the serotypes contained in V116 was determined using a multiplex opsonophagocytic assay (MOPA). Geometric mean fold rise (GMFR) is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline. The GMFRs in OPA responses from baseline to 30 days post-vaccination with 95% confidence intervals are presented.
Time Frame: Day 1 (Baseline) and 30 days post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 212 | 115 | 164 | 76 | 98
Ratio
  Serotype 3: number analyzed (Participants) | 164 | 91 | 131 | 68 | 76
  Serotype 3 | 4.4 [3.7 to 5.3] | 4.0 [3.1 to 5.3] | 6.2 [5.0 to 7.6] | 7.5 [5.3 to 10.5] | 5.0 [3.6 to 7.0]
  Serotype 6A: number analyzed (Participants) | 171 | 87 | 136 | 66 | 89
  Serotype 6A | 6.2 [5.0 to 7.7] | 7.1 [4.9 to 10.3] | 4.2 [3.3 to 5.3] | 1.8 [1.4 to 2.4] | 5.5 [4.1 to 7.4]
  Serotype 7F: number analyzed (Participants) | 200 | 102 | 146 | 69 | 92
  Serotype 7F | 4.1 [3.3 to 5.1] | 3.9 [2.8 to 5.4] | 4.6 [3.6 to 5.9] | 4.2 [3.1 to 5.8] | 3.9 [2.9 to 5.3]
  Serotype 19A: number analyzed (Participants) | 194 | 104 | 149 | 72 | 90
  Serotype 19A | 2.4 [2.0 to 2.8] | 3.3 [2.5 to 4.4] | 2.8 [2.3 to 3.3] | 3.6 [2.7 to 4.7] | 2.5 [1.8 to 3.3]
  Serotype 22F: number analyzed (Participants) | 193 | 102 | 124 | 64 | 94
  Serotype 22F | 7.0 [5.5 to 9.0] | 7.1 [4.8 to 10.6] | 26.3 [17.7 to 39.2] | 14.8 [8.7 to 25.1] | 7.5 [4.9 to 11.4]
  Serotype 33F: number analyzed (Participants) | 177 | 93 | 125 | 50 | 85
  Serotype 33F | 2.2 [1.8 to 2.6] | 1.7 [1.3 to 2.4] | 6.3 [4.8 to 8.4] | 9.2 [5.6 to 15.3] | 2.7 [2.0 to 3.7]
  Serotype 8: number analyzed (Participants) | 198 | 108 | 151 | 71 | 96
  Serotype 8 | 2.8 [2.4 to 3.4] | 0.9 [0.7 to 1.0] | 16.6 [12.2 to 22.7] | 18.6 [11.9 to 29.1] | 3.8 [2.7 to 5.3]
  Serotype 9N: number analyzed (Participants) | 186 | 108 | 136 | 53 | 87
  Serotype 9N | 2.3 [2.0 to 2.7] | 1.4 [1.1 to 1.7] | 5.9 [4.7 to 7.4] | 6.8 [4.7 to 9.8] | 3.5 [2.7 to 4.5]
  Serotype 10A: number analyzed (Participants) | 200 | 111 | 148 | 71 | 93
  Serotype 10A | 4.3 [3.5 to 5.4] | 1.0 [0.9 to 1.2] | 17.1 [12.7 to 23.0] | 11.8 [7.5 to 18.6] | 4.7 [3.4 to 6.5]
  Serotype 11A: number analyzed (Participants) | 186 | 91 | 131 | 65 | 83
  Serotype 11A | 6.5 [5.2 to 8.2] | 1.2 [0.9 to 1.7] | 21.0 [14.6 to 30.4] | 9.2 [5.9 to 14.4] | 9.5 [6.2 to 14.4]
  Serotype 12F: number analyzed (Participants) | 207 | 112 | 157 | 72 | 93
  Serotype 12F | 11.8 [9.0 to 15.4] | 1.1 [1.0 to 1.3] | 82.2 [62.9 to 107.4] | 41.9 [26.1 to 67.2] | 13.7 [9.0 to 20.8]
  Serotype 15A: number analyzed (Participants) | 142 | 78 | 110 | 40 | 62
  Serotype 15A | 5.6 [4.3 to 7.4] | 1.2 [0.9 to 1.5] | 9.0 [6.8 to 11.8] | 3.0 [2.0 to 4.5] | 7.2 [4.6 to 11.2]
  Serotype 15C: number analyzed (Participants) | 197 | 108 | 141 | 68 | 82
  Serotype 15C | 8.5 [6.7 to 10.9] | 1.3 [1.0 to 1.7] | 30.6 [22.5 to 41.5] | 12.7 [8.5 to 18.8] | 11.6 [8.1 to 16.4]
  Serotype 16F: number analyzed (Participants) | 172 | 100 | 132 | 68 | 86
  Serotype 16F | 7.1 [5.9 to 8.5] | 1.1 [0.9 to 1.3] | 9.8 [7.8 to 12.4] | 2.0 [1.5 to 2.7] | 7.2 [5.5 to 9.6]
  Serotype 17F: number analyzed (Participants) | 183 | 101 | 116 | 64 | 79
  Serotype 17F | 3.7 [3.0 to 4.5] | 0.9 [0.8 to 1.1] | 13.5 [9.5 to 19.2] | 8.1 [5.6 to 11.7] | 6.5 [4.6 to 9.3]
  Serotype 20A: number analyzed (Participants) | 184 | 105 | 129 | 69 | 81
  Serotype 20A | 3.7 [3.0 to 4.5] | 0.9 [0.8 to 1.0] | 12.2 [9.3 to 16.0] | 6.0 [4.4 to 8.3] | 4.4 [3.1 to 6.1]
  Serotype 23A: number analyzed (Participants) | 157 | 76 | 118 | 38 | 65
  Serotype 23A | 8.4 [6.2 to 11.6] | 1.4 [1.0 to 1.9] | 19.0 [13.5 to 26.9] | 2.5 [1.3 to 4.9] | 16.3 [10.3 to 25.7]
  Serotype 23B: number analyzed (Participants) | 191 | 109 | 155 | 71 | 94
  Serotype 23B | 21.4 [16.2 to 28.1] | 4.2 [2.9 to 6.0] | 35.5 [25.9 to 48.6] | 5.2 [3.5 to 7.6] | 26.1 [17.5 to 38.9]
  Serotype 24F: number analyzed (Participants) | 187 | 91 | 127 | 61 | 82
  Serotype 24F | 25.8 [19.5 to 34.0] | 1.0 [0.8 to 1.3] | 31.1 [22.8 to 42.6] | 0.9 [0.7 to 1.3] | 39.5 [27.4 to 56.9]
  Serotype 31: number analyzed (Participants) | 179 | 97 | 134 | 61 | 84
  Serotype 31 | 16.7 [12.5 to 22.3] | 0.9 [0.7 to 1.2] | 35.6 [24.8 to 51.2] | 1.7 [1.1 to 2.6] | 30.5 [19.1 to 48.6]
  Serotype 35B: number analyzed (Participants) | 183 | 106 | 144 | 71 | 85
  Serotype 35B | 6.0 [4.8 to 7.4] | 1.0 [0.8 to 1.2] | 7.2 [5.6 to 9.2] | 1.4 [1.1 to 1.8] | 5.7 [4.2 to 7.9]

7. Secondary Outcome: Percentage of Participants Who Achieve a ≥4-fold Increase in Serotype-specific OPA Responses
Description: Activity for the serotypes contained in V116 was determined using a MOPA. The percentage of participants with a ≥4-fold rise from baseline to at 30 days post-vaccination for OPA responses with 95% confidence intervals are presented.
Time Frame: Day 1 (Baseline) and 30 days post-vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 212 | 115 | 164 | 76 | 98
Percentage of Participants
  Serotype 3: number analyzed (Participants) | 164 | 91 | 131 | 68 | 76
  Serotype 3 | 54.9 [46.9 to 62.6] | 54.9 [44.2 to 65.4] | 64.1 [55.3 to 72.3] | 66.2 [53.7 to 77.2] | 48.7 [37.0 to 60.4]
  Serotype 6A: number analyzed (Participants) | 171 | 87 | 136 | 66 | 89
  Serotype 6A | 57.9 [50.1 to 65.4] | 58.6 [47.6 to 69.1] | 46.3 [37.7 to 55.1] | 18.2 [9.8 to 29.6] | 56.2 [45.3 to 66.7]
  Serotype 7F: number analyzed (Participants) | 200 | 102 | 146 | 69 | 92
  Serotype 7F | 38.5 [31.7 to 45.6] | 43.1 [33.4 to 53.3] | 44.5 [36.3 to 53.0] | 49.3 [37.0 to 61.6] | 38.0 [28.1 to 48.8]
  Serotype 19A: number analyzed (Participants) | 194 | 104 | 149 | 72 | 90
  Serotype 19A | 28.4 [22.1 to 35.2] | 34.6 [25.6 to 44.6] | 33.6 [26.0 to 41.7] | 38.9 [27.6 to 51.1] | 30.0 [20.8 to 40.6]
  Serotype 22F: number analyzed (Participants) | 193 | 102 | 124 | 64 | 94
  Serotype 22F | 53.9 [46.6 to 61.1] | 54.9 [44.7 to 64.8] | 77.4 [69.0 to 84.4] | 65.6 [52.7 to 77.1] | 50.0 [39.5 to 60.5]
  Serotype 33F: number analyzed (Participants) | 177 | 93 | 125 | 50 | 85
  Serotype 33F | 19.8 [14.2 to 26.4] | 19.4 [11.9 to 28.9] | 52.0 [42.9 to 61.0] | 56.0 [41.3 to 70.0] | 29.4 [20.0 to 40.3]
  Serotype 8: number analyzed (Participants) | 198 | 108 | 151 | 71 | 96
  Serotype 8 | 33.3 [26.8 to 40.4] | 2.8 [0.6 to 7.9] | 70.2 [62.2 to 77.4] | 74.6 [62.9 to 84.2] | 34.4 [25.0 to 44.8]
  Serotype 9N: number analyzed (Participants) | 186 | 108 | 136 | 53 | 87
  Serotype 9N | 22.0 [16.3 to 28.7] | 6.5 [2.6 to 12.9] | 57.4 [48.6 to 65.8] | 67.9 [53.7 to 80.1] | 39.1 [28.8 to 50.1]
  Serotype 10A: number analyzed (Participants) | 200 | 111 | 148 | 71 | 93
  Serotype 10A | 46.0 [38.9 to 53.2] | 2.7 [0.6 to 7.7] | 74.3 [66.5 to 81.1] | 67.6 [55.5 to 78.2] | 49.5 [38.9 to 60.0]
  Serotype 11A: number analyzed (Participants) | 186 | 91 | 131 | 65 | 83
  Serotype 11A | 53.8 [46.3 to 61.1] | 12.1 [6.2 to 20.6] | 73.3 [64.8 to 80.6] | 53.8 [41.0 to 66.3] | 59.0 [47.7 to 69.7]
  Serotype 12F: number analyzed (Participants) | 207 | 112 | 157 | 72 | 93
  Serotype 12F | 62.8 [55.8 to 69.4] | 6.3 [2.5 to 12.5] | 93.0 [87.8 to 96.5] | 81.9 [71.1 to 90.0] | 60.2 [49.5 to 70.2]
  Serotype 15A: number analyzed (Participants) | 142 | 78 | 110 | 40 | 62
  Serotype 15A | 53.5 [45.0 to 61.9] | 12.8 [6.3 to 22.3] | 70.9 [61.5 to 79.2] | 35.0 [20.6 to 51.7] | 59.7 [46.4 to 71.9]
  Serotype 15C: number analyzed (Participants) | 197 | 108 | 141 | 68 | 82
  Serotype 15C | 61.4 [54.2 to 68.3] | 10.2 [5.2 to 17.5] | 84.4 [77.3 to 90.0] | 72.1 [59.9 to 82.3] | 72.0 [60.9 to 81.3]
  Serotype 16F: number analyzed (Participants) | 172 | 100 | 132 | 68 | 86
  Serotype 16F | 68.0 [60.5 to 74.9] | 8.0 [3.5 to 15.2] | 70.5 [61.9 to 78.1] | 30.9 [20.2 to 43.3] | 70.9 [60.1 to 80.2]
  Serotype 17F: number analyzed (Participants) | 183 | 101 | 116 | 64 | 79
  Serotype 17F | 37.7 [30.7 to 45.2] | 2.0 [0.2 to 7.0] | 74.1 [65.2 to 81.8] | 62.5 [49.5 to 74.3] | 54.4 [42.8 to 65.7]
  Serotype 20A: number analyzed (Participants) | 184 | 105 | 129 | 69 | 81
  Serotype 20A | 37.5 [30.5 to 44.9] | 2.9 [0.6 to 8.1] | 76.7 [68.5 to 83.7] | 60.9 [48.4 to 72.4] | 46.9 [35.7 to 58.3]
  Serotype 23A: number analyzed (Participants) | 157 | 76 | 118 | 38 | 65
  Serotype 23A | 59.9 [51.8 to 67.6] | 21.1 [12.5 to 31.9] | 73.7 [64.8 to 81.4] | 34.2 [19.6 to 51.4] | 80.0 [68.2 to 88.9]
  Serotype 23B: number analyzed (Participants) | 191 | 109 | 155 | 71 | 94
  Serotype 23B | 74.9 [68.1 to 80.9] | 40.4 [31.1 to 50.2] | 80.6 [73.5 to 86.5] | 43.7 [31.9 to 56.0] | 80.9 [71.4 to 88.2]
  Serotype 24F: number analyzed (Participants) | 187 | 91 | 127 | 61 | 82
  Serotype 24F | 80.2 [73.8 to 85.7] | 7.7 [3.1 to 15.2] | 81.9 [74.1 to 88.2] | 4.9 [1.0 to 13.7] | 89.0 [80.2 to 94.9]
  Serotype 31: number analyzed (Participants) | 179 | 97 | 134 | 61 | 84
  Serotype 31 | 70.9 [63.7 to 77.5] | 8.2 [3.6 to 15.6] | 81.3 [73.7 to 87.5] | 18.0 [9.4 to 30.0] | 82.1 [72.3 to 89.6]
  Serotype 35B: number analyzed (Participants) | 183 | 106 | 144 | 71 | 85
  Serotype 35B | 55.2 [47.7 to 62.5] | 7.5 [3.3 to 14.3] | 65.3 [56.9 to 73.0] | 7.0 [2.3 to 15.7] | 57.6 [46.4 to 68.3]

8. Secondary Outcome: Geometric Mean Fold Rise of Serotype-specific IgG
Description: Activity for the serotypes contained in V116 was determined using a PnECL assay. Geometric mean fold rise (GMFR) is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline. The GMFRs IgG responses from baseline to 30 days post-vaccination with 95% confidence intervals are presented.
Time Frame: Day 1 (Baseline) and 30 days post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 220 | 117 | 167 | 81 | 99
Ratio
  Serotype 3 | 3.6 [3.2 to 4.0] | 3.1 [2.6 to 3.7] | 3.7 [3.2 to 4.3] | 5.7 [4.3 to 7.4] | 2.9 [2.3 to 3.5]
  Serotype 6A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 6A | 5.9 [5.0 to 7.1] | 8.0 [6.1 to 10.6] | 3.3 [2.7 to 4.0] | 2.5 [1.9 to 3.2] | 4.4 [3.4 to 5.7]
  Serotype 7F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 7F | 3.3 [2.8 to 3.8] | 2.9 [2.3 to 3.5] | 3.2 [2.7 to 3.8] | 3.2 [2.6 to 3.9] | 3.2 [2.6 to 4.0]
  Serotype 19A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 19A | 2.3 [2.0 to 2.7] | 3.4 [2.8 to 4.2] | 2.2 [1.9 to 2.5] | 3.0 [2.4 to 3.6] | 2.0 [1.7 to 2.4]
  Serotype 22F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 22F | 4.2 [3.6 to 4.9] | 3.4 [2.8 to 4.2] | 14.3 [11.4 to 18.0] | 8.5 [6.2 to 11.6] | 3.5 [2.7 to 4.6]
  Serotype 33F | 2.2 [1.9 to 2.5] | 1.8 [1.5 to 2.1] | 8.6 [7.1 to 10.5] | 10.5 [7.9 to 13.9] | 2.4 [1.9 to 3.0]
  Serotype 8 | 2.7 [2.4 to 3.1] | 1.0 [0.9 to 1.1] | 12.1 [9.8 to 15.0] | 14.4 [10.3 to 20.0] | 2.3 [1.9 to 2.8]
  Serotype 9N: number analyzed (Participants) | 217 | 117 | 167 | 81 | 99
  Serotype 9N | 2.9 [2.4 to 3.4] | 1.4 [1.2 to 1.6] | 8.7 [7.1 to 10.6] | 9.1 [6.8 to 12.1] | 3.2 [2.6 to 3.9]
  Serotype 10A | 4.4 [3.7 to 5.2] | 1.0 [0.9 to 1.0] | 18.9 [15.3 to 23.4] | 10.1 [7.6 to 13.4] | 4.2 [3.1 to 5.5]
  Serotype 11A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 11A | 4.1 [3.6 to 4.7] | 1.0 [0.9 to 1.0] | 10.3 [8.5 to 12.6] | 5.6 [4.4 to 7.2] | 3.5 [2.7 to 4.3]
  Serotype 12F | 4.2 [3.6 to 5.0] | 1.0 [0.9 to 1.1] | 14.2 [11.3 to 17.9] | 8.4 [5.8 to 12.0] | 3.5 [2.7 to 4.5]
  Serotype 15A | 12.2 [10.1 to 14.7] | 1.0 [0.9 to 1.1] | 24.5 [19.7 to 30.3] | 2.4 [2.0 to 3.0] | 16.6 [12.0 to 22.9]
  Serotype 15C: number analyzed (Participants) | 219 | 117 | 166 | 81 | 99
  Serotype 15C | 5.8 [4.9 to 6.9] | 1.0 [0.9 to 1.2] | 18.8 [14.9 to 23.8] | 6.2 [4.8 to 8.2] | 6.4 [5.0 to 8.1]
  Serotype 16F: number analyzed (Participants) | 218 | 117 | 166 | 81 | 99
  Serotype 16F | 15.2 [12.7 to 18.2] | 1.1 [1.0 to 1.2] | 15.7 [12.9 to 19.0] | 1.6 [1.3 to 1.8] | 11.9 [9.2 to 15.4]
  Serotype 17F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 17F | 4.7 [4.0 to 5.5] | 1.0 [0.9 to 1.1] | 17.4 [14.3 to 21.1] | 10.5 [7.8 to 14.1] | 3.8 [2.9 to 5.0]
  Serotype 20A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 20A | 3.8 [3.3 to 4.4] | 1.0 [0.9 to 1.1] | 14.8 [12.2 to 17.9] | 8.5 [6.4 to 11.4] | 3.7 [2.9 to 4.8]
  Serotype 23A: number analyzed (Participants) | 219 | 117 | 166 | 81 | 99
  Serotype 23A | 13.5 [11.1 to 16.5] | 1.8 [1.5 to 2.2] | 18.9 [15.3 to 23.4] | 2.3 [1.9 to 2.7] | 13.1 [9.6 to 17.7]
  Serotype 23B: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 23B | 8.2 [6.7 to 10.0] | 2.7 [2.1 to 3.5] | 7.3 [6.0 to 8.9] | 2.3 [1.9 to 2.9] | 7.3 [5.4 to 9.7]
  Serotype 24F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 24F | 26.9 [21.8 to 33.1] | 1.0 [0.9 to 1.1] | 21.7 [17.3 to 27.2] | 1.0 [0.9 to 1.1] | 24.4 [17.1 to 34.9]
  Serotype 31: number analyzed (Participants) | 217 | 117 | 167 | 81 | 90
  Serotype 31 | 13.1 [11.0 to 15.6] | 1.1 [1.0 to 1.2] | 14.4 [11.9 to 17.3] | 1.5 [1.3 to 1.8] | 13.0 [9.9 to 17.0]
  Serotype 35B: number analyzed (Participants) | 218 | 117 | 167 | 81 | 99
  Serotype 35B | 16.8 [13.9 to 20.3] | 1.0 [0.9 to 1.0] | 15.6 [12.9 to 18.7] | 0.9 [0.9 to 1.0] | 15.7 [11.9 to 20.8]

9. Secondary Outcome: Percentage of Participants Who Achieve a ≥4-fold Increase in Serotype-specific IgG Response
Description: Activity for the serotypes contained in V116 was determined using a PnECL assay. The percentage of participants with a ≥4-fold rise from baseline to at 30 days post-vaccination for IgG responses with 95% confidence intervals are presented.
Time Frame: Day 1 (Baseline) and 30 days post-vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
Number analyzed (Participants) | 220 | 117 | 167 | 81 | 99
Percentage of Participants
  Serotype 3 | 42.7 [36.1 to 49.6] | 36.8 [28.0 to 46.2] | 40.7 [33.2 to 48.6] | 54.3 [42.9 to 65.4] | 35.4 [26.0 to 45.6]
  Serotype 6A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 6A | 56.2 [49.3 to 62.8] | 65.0 [55.6 to 73.5] | 35.9 [28.7 to 43.7] | 27.2 [17.9 to 38.2] | 45.5 [35.4 to 55.8]
  Serotype 7F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 7F | 34.7 [28.4 to 41.4] | 29.9 [21.8 to 39.1] | 37.7 [30.4 to 45.5] | 33.3 [23.2 to 44.7] | 37.4 [27.9 to 47.7]
  Serotype 19A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 19A | 24.7 [19.1 to 30.9] | 37.6 [28.8 to 47.0] | 19.8 [14.0 to 26.6] | 33.3 [23.2 to 44.7] | 19.2 [12.0 to 28.3]
  Serotype 22F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 22F | 39.3 [32.8 to 46.1] | 35.0 [26.5 to 44.4] | 78.4 [71.4 to 84.4] | 65.4 [54.0 to 75.7] | 43.4 [33.5 to 53.8]
  Serotype 33F | 19.1 [14.1 to 24.9] | 12.8 [7.4 to 20.3] | 72.5 [65.0 to 79.1] | 75.3 [64.5 to 84.2] | 27.3 [18.8 to 37.1]
  Serotype 8 | 29.5 [23.6 to 36.0] | 0.9 [0.0 to 4.7] | 78.4 [71.4 to 84.4] | 76.5 [65.8 to 85.2] | 26.3 [17.9 to 36.1]
  Serotype 9N: number analyzed (Participants) | 217 | 117 | 167 | 81 | 99
  Serotype 9N | 31.8 [25.7 to 38.4] | 7.7 [3.6 to 14.1] | 68.9 [61.2 to 75.8] | 72.8 [61.8 to 82.1] | 36.4 [26.9 to 46.6]
  Serotype 10A | 45.5 [38.7 to 52.3] | 0.9 [0.0 to 4.7] | 82.6 [76.0 to 88.1] | 80.2 [69.9 to 88.3] | 46.5 [36.4 to 56.8]
  Serotype 11A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 11A | 43.8 [37.2 to 50.7] | 0.0 [0.0 to 3.1] | 72.5 [65.0 to 79.1] | 63.0 [51.5 to 73.4] | 43.4 [33.5 to 53.8]
  Serotype 12F | 44.5 [37.9 to 51.4] | 2.6 [0.5 to 7.3] | 75.4 [68.2 to 81.8] | 60.5 [49.0 to 71.2] | 39.4 [29.7 to 49.7]
  Serotype 15A | 73.6 [67.3 to 79.3] | 0.9 [0.0 to 4.7] | 89.8 [84.2 to 94.0] | 28.4 [18.9 to 39.5] | 77.8 [68.3 to 85.5]
  Serotype 15C: number analyzed (Participants) | 219 | 117 | 166 | 81 | 99
  Serotype 15C | 57.5 [50.7 to 64.2] | 3.4 [0.9 to 8.5] | 80.1 [73.2 to 85.9] | 64.2 [52.8 to 74.6] | 66.7 [56.5 to 75.8]
  Serotype 16F: number analyzed (Participants) | 218 | 117 | 166 | 81 | 99
  Serotype 16F | 82.1 [76.4 to 87.0] | 2.6 [0.5 to 7.3] | 84.9 [78.6 to 90.0] | 13.6 [7.0 to 23.0] | 77.8 [68.3 to 85.5]
  Serotype 17F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 17F | 48.9 [42.1 to 55.7] | 1.7 [0.2 to 6.0] | 83.8 [77.4 to 89.1] | 74.1 [63.1 to 83.2] | 44.4 [34.5 to 54.8]
  Serotype 20A: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 20A | 36.5 [30.1 to 43.3] | 0.9 [0.0 to 4.7] | 83.2 [76.7 to 88.6] | 69.1 [57.9 to 78.9] | 49.5 [39.3 to 59.7]
  Serotype 23A: number analyzed (Participants) | 219 | 117 | 166 | 81 | 99
  Serotype 23A | 77.6 [71.5 to 83.0] | 17.1 [10.8 to 25.2] | 86.7 [80.6 to 91.5] | 21.0 [12.7 to 31.5] | 77.8 [68.3 to 85.5]
  Serotype 23B: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 23B | 64.8 [58.1 to 71.2] | 26.5 [18.8 to 35.5] | 60.5 [52.6 to 67.9] | 21.0 [12.7 to 31.5] | 64.6 [54.4 to 74.0]
  Serotype 24F: number analyzed (Participants) | 219 | 117 | 167 | 81 | 99
  Serotype 24F | 85.4 [80.0 to 89.8] | 0.0 [0.0 to 3.1] | 88.0 [82.1 to 92.5] | 0.0 [0.0 to 4.5] | 83.8 [75.1 to 90.5]
  Serotype 31: number analyzed (Participants) | 217 | 117 | 167 | 81 | 99
  Serotype 31 | 79.7 [73.8 to 84.9] | 2.6 [0.5 to 7.3] | 84.4 [78.0 to 89.6] | 11.1 [5.2 to 20.0] | 80.8 [71.7 to 88.0]
  Serotype 35B: number analyzed (Participants) | 218 | 117 | 167 | 81 | 99
  Serotype 35B | 83.9 [78.4 to 88.6] | 0.0 [0.0 to 3.1] | 82.6 [76.0 to 88.1] | 0.0 [0.0 to 4.5] | 84.8 [76.2 to 91.3]

ADVERSE EVENTS:
Time Frame: Up to approximately 30 days post-vaccination for non-serious adverse events (AEs) and up to approximately 180 days for serious AEs and deaths.
Description: The analysis population for All-Cause Mortality included all randomized participants. The safety analysis population included all randomized participants who received the study vaccination.
Arm/Group | Cohort 1: V116 | Cohort 1: PCV15 | Cohort 2: V116 | Cohort 2: PPSV23 | Cohort 3: V116
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/119 | 0/176 | 0/85 | 0/106
Serious Adverse Events (participants affected / at risk) | 2/230 | 4/117 | 2/174 | 3/85 | 2/105
Other Adverse Events (participants affected / at risk) | 107/230 | 66/117 | 85/174 | 52/85 | 51/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: V116 (N=230) | Cohort 1: PCV15 (N=117) | Cohort 2: V116 (N=174) | Cohort 2: PPSV23 (N=85) | Cohort 3: V116 (N=105)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortoenteric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: V116 (N=230) | Cohort 1: PCV15 (N=117) | Cohort 2: V116 (N=174) | Cohort 2: PPSV23 (N=85) | Cohort 3: V116 (N=105)
Fatigue (General disorders) | 33 (33) | 20 (20) | 33 (34) | 12 (12) | 23 (23)
Injection site erythema (General disorders) | 19 (19) | 9 (9) | 14 (14) | 8 (8) | 8 (8)
Injection site pain (General disorders) | 82 (82) | 51 (51) | 72 (72) | 40 (40) | 46 (46)
Injection site swelling (General disorders) | 20 (20) | 10 (10) | 8 (8) | 14 (14) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 5 (5) | 17 (17) | 9 (9) | 9 (9)
Headache (Nervous system disorders) | 17 (17) | 11 (11) | 18 (19) | 10 (10) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT05420961/Prot_SAP_000.pdf